CLINICAL TRIAL: NCT00415363
Title: A Double-blind, Randomized, Placebo-controlled Multicentre Phase II Study of Maintenance Enzastaurin Following Whole Brain Radiation Therapy in the Treatment of Brain Metastases From Lung Cancer
Brief Title: Study of Enzastaurin Versus Placebo in the Treatment of Patients With Brain Metastases of Lung Cancer, After Whole Brain Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10710; H6Q-MC-S020 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — enzastaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: enzastaurin
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily, until disease progression
  Other Names: LY317615
  Arms: A
Drug: placebo — oral, daily
  Arms: B

SUMMARY:
This study is a multinational study to compare enzastaurin versus placebo in the treatment of patients with brain metastases of lung cancer. Approximately 108 patients will be randomly assigned to receive either enzastaurin or placebo after having completed whole brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Having radiologically proven brain metastases of lung cancer
* Having received whole brain radiotherapy with either 30 grays in 2 weeks or 20 grays in one week. Treatment with enzastaurin must start within 14 days after the last fraction of the whole brain radiotherapy
* No other previous radiotherapy to the brain except for radiosurgery at one occasion
* Adequate organ function as measured by appropriate laboratory tests.
* Age 18 years or older.

Exclusion Criteria:

* Inability to swallow tablets or show conditions which could interfere with oral medication intake (e.g. vomiting, partial bowel obstruction).
* Inability to discontinue use of certain anti-epileptic drugs such as, carbamazepine, phenobarbital or phenytoin.
* Concurrent administration of warfarin
* Hemophilia
* Having had any systemic anti-cancer treatment within the last 2 weeks prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours,, EST), Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen, Denmark
- Norway (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trondheim
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn, Poland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca, Romania
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzastaurin: Enzastaurin delivered as 1125 mg loading dose then 500 mg, oral, daily, until disease progression
- Placebo: Placebo delivered as identical in appearance oral dose, daily.
Period: Overall Study
Arm/Group | Enzastaurin | Placebo
Started | 55 | 54
Safety Population | 54 | 53
Completed | 0 | 0
Not Completed | 55 | 54
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Death | 16 | 12
Not completed — Progressive disease | 26 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzastaurin | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (7.4) | 63.5 (10.0) | 63.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 31 | 34 | 65
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 0 | 2 | 2
  Romania | 15 | 13 | 28
  Denmark | 4 | 2 | 6
  Norway | 26 | 28 | 54
  Sweden | 6 | 7 | 13
  Finland | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression of Brain Metastases
Description: Time to progression (TTP) of brain metastases is the time from randomization to first observation of brain metastases progression. Response Evaluation Criteria In Solid Tumors (RECIST; Version 1.0), using magnetic resonance imaging (MRI), until observation of objective progression, or clinically as the date of increased steroids dose (barring radiological confirmation), was used to assess progressive disease (PD) of brain metastases. TTP was right-censored with the date of last contact if the participant died without MRI-documented PD or symptomatic deterioration or was lost to follow-up or received post therapy (Radio, Systemic, Surgery) before documented PD of the brain metastases.
Time Frame: Baseline to measured progressive disease (up to 21.2 months)
Population: Time to progressive disease (TTP) was analyzed on all randomized patients. Participants censored: Enzastaurin = 35 and Placebo = 32.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 55 | 54
months | 6.9 [3.4 to 11.9] | 4.9 [3.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Time to Objective Progression of Brain Metastases
Description: Time to objective progression (TTOP) of brain metastases is the time from randomization to the first observation of objective progression of brain metastases assessed by MRI.
  TTOP was right-censored with the date of the last objective progression-free disease assessment if the participant died or did not have objective PD as of the cut-off date. For participants receiving post-discontinuation therapy prior to PD of brain metastases, TTOP was censored at the last assessment before post-discontinuation therapy. Kaplan-Meier estimated the median survival times and confidence intervals.
Time Frame: Baseline to measured progressive disease (up to 21.2 months)
Population: TTOP was analyzed on randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 55 | 54
months | 5.0 [3.1 to 8.4] | 3.7 [3.4 to 8.2]

3. Secondary Outcome: Overall Progression-free Survival (Including Both Progression of Brain and Extracranial Tumor Lesion)
Description: Overall progression-free survival (PFS) is defined as the time from the date of study enrollment to the first date of progressive disease or death from any cause.
  For participants not known to have died as of the data cut-off date and who did not have progressive disease, PFS was censored at last contact date. For those who received subsequent systemic anticancer therapy (after discontinuation from study therapy) prior to objectively determined progression of brain metastases, PFS was censored at the start of radiotherapy for extracranial lesions or the date of starting chemotherapy.
Time Frame: Baseline to measured progressive disease (up to 14.4 months)
Population: Progression-free survival was analyzed on all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 55 | 54
months | 2.2 [1.1 to 2.3] | 2.0 [1.3 to 2.3]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS was censored at the last contact date.
Time Frame: Baseline to date of death from any cause (up to 27.2 months)
Population: OS was analyzed on all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 55 | 54
months | 3.8 [2.6 to 5.6] | 5.1 [3.7 to 5.7]

5. Secondary Outcome: Overall Response (OR) to Treatment of Extra-cranial Tumor Lesions by Percentage of Participants
Description: Overall Response (OR) was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST v1.0). OR on extra-cranial tumors was assessed by response sequences. Complete response (CR) or partial response (PR), was confirmed by second assessment performed >= 28 days after first response. Two CRs before progression required for best response of CR. Two PRs or better not qualifying for a CR, for best response of PR.
  * CR: Disappearance of all tumor lesions.
  * PR: 30% decrease from baseline in sum of the longest diameter of target lesions or complete disappearance of target lesions, without worsening of one or more nontarget lesions. In either case, no new lesions may have appeared.
  * Stable Disease (SD) is defined as disease that does not meet the criteria for CR, PR, or progressive disease (PD), and has been evaluated at least 1 time, at least 6 weeks after baseline assessment.
Time Frame: Baseline to measured progressive disease (up to 27.2 months)
Population: Rate and 95% confidence intervals of overall response to treatment of extra-cranial tumor lesions were evaluated on all randomized participants who qualified for tumor response analysis by the following criteria:
  * Presence of measurable disease in at least one site other than brain
  * Treatment with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 41 | 44
percentage of participants
  Complete Response | 0 [0 to 8.6] | 0 [0 to 15.5]
  Partial Response | 0 [0 to 8.6] | 4.5 [0.6 to 15.5]
  Stable Disease | 12.2 [4.1 to 26.2] | 25.0 [13.2 to 40.3]
  Progressive Disease | 58.5 [42.1 to 73.7] | 47.7 [32.5 to 63.3]
  Unknown/Not Done | 29.3 [16.1 to 45.5] | 22.7 [11.5 to 37.8]

6. Secondary Outcome: Best Overall Tumor Response on Brain Metastases by Percentage of Participants
Description: Best overall tumor response on brain metastases (BOR) according to RECIST V1.0 response criteria. For complete response (CR) or partial response (PR), BOR was to be confirmed. Response criteria were
  * CR: Disappearance of all tumor lesions.
  * PR: Either a) at least a 30% decrease in sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LDs or b) complete disappearance of target lesions, with persistence (but not worsening) of one or more nontarget lesions. In either case, no new lesions may have appeared.
  * Stable Disease (SD) is defined as disease that does not meet the criteria for CR, PR, or progressive disease (PD), and has been evaluated at least 1 time, at least 6 weeks after baseline assessment.
Time Frame: Baseline to measured progressive disease (up to 21.2 months)
Population: Best overall tumor response (BOR) on brain metastases and 95% confidence intervals were evaluated on all randomized patients who qualified by the following criteria:
  * Presence of measurable disease in brain
  * Treatment with at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 43 | 44
percentage of participants
  Complete Response | 0 [0 to 8.2] | 2.3 [0.1 to 12.0]
  Partial Response | 9.3 [2.6 to 22.1] | 4.5 [0.6 to 15.5]
  Stable Disease | 34.9 [21.0 to 50.9] | 50 [34.6 to 65.4]
  Progressive Disease | 14.0 [5.3 to 27.9] | 18.2 [8.2 to 32.7]
  Unknown/Not Done | 41.9 [27.0 to 57.9] | 25.0 [13.2 to 40.3]

7. Secondary Outcome: Health-related Quality of Life (HRQoL) EORTC QLQ-C30 Physical Functioning
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). Physical functioning was measured by items 1 to 5. Their sum score was linearly transformed to the range 0 - 100 as recommended by the EORTC (higher score is better).
Time Frame: Baseline to 30 days after discontinuation (up to 17.6 months)
Population: EORTC QLQ-C30 scores from all randomized patients who filled in at least baseline and one post baseline questionnaire were evaluated and summarized by means of descriptive statistics.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 42 | 43
units on a scale
  Week 3 | -6.7 [-20.0 to 0] | -8.3 [-20.0 to 0]
  Week 6 | -20.0 [-40.0 to 0] | -13.3 [-30.0 to 6.7]
  Week 9 | -13.3 [-46.7 to -6.7] | -13.3 [-30.0 to -6.7]
  Week 12 | -13.3 [-13.3 to 5.0] | -26.7 [-46.7 to -6.7]
  Week 15 | 6.7 [-6.7 to 20.0] | -13.3 [-26.7 to 0]
  Week 18 | 20.0 [20.0 to 20.0] | -30.0 [-40.0 to -6.7]
  Week 21 | 0 [0 to 0] | 13.3 [0 to 13.3]
  Week 24 | 20.0 [20.0 to 20.0] | 13.3 [13.3 to 13.3]
  Week 27 | 0 [0 to 0] | 0 [0 to 0]
  Week 30 | 0 [0 to 0] | -60.0 [-60.0 to -60.0]
  Week 33 | 0 [0 to 0] | -73.3 [-73.3 to -73.3]
  30 days post last therapy | -13.3 [-40.0 to 0] | -20.0 [-46.7 to -13.3]

8. Secondary Outcome: HRQoL Questionnaire - EORTC QLQ-C30 Fatigue
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100 (lower score is better).
Time Frame: Baseline to 30 days after discontinuation (up to 17.6 months)
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 42 | 43
units on a scale
  Week 4 | 0 [0 to 22.2] | 0 [0 to 22.2]
  Week 7 | 22.2 [0 to 38.9] | 0 [-11.1 to 22.2]
  Week 10 | 11.1 [-22.2 to 22.2] | 5.6 [-16.7 to 33.3]
  Week 13 | 0 [-11.1 to 22.2] | 0 [-11.1 to 33.3]
  Week 16 | 5.6 [-11.1 to 22.2] | 0 [-11.1 to 22.2]
  Week 19 | 11.1 [11.1 to 11.1] | 11.1 [-5.6 to 16.7]
  Week 22 | 0 [0 to 0] | 0 [-11.1 to 11.1]
  Week 25 | 22.2 [22.2 to 22.2] | -11.1 [-11.1 to -11.1]
  Week 28 | 0 [0 to 0] | 0 [0 to 0]
  Week 31 | 0 [0 to 0] | 55.6 [55.6 to 55.6]
  Week 34 | 0 [0 to 0] | 77.8 [77.8 to 77.8]
  30 days post last therapy | 0 [-11.1 to 11.1] | 22.2 [0 to 55.6]

9. Secondary Outcome: HRQoL Questionnaire - EORTC QLQ-C30 Nausea/Vomiting
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Nausea/Vomiting Scale is scored between 0 and 100 (lower score is better).
Time Frame: Baseline to 30 days after discontinuation (up to 17.6 months)
Population: EORTC QLQ-C30 scores from all randomized patients who filled in at least baseline and one post baseline questionnaire were evaluated and summarized by means of descriptive statistics. Median differences between treatment groups in change from baseline to every 4 weeks and the inter-quartile range are reported.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 42 | 43
units on a scale
  Week 4 | 0 [-16.7 to 16.7] | 0 [0 to 0]
  Week 7 | 0 [-16.7 to 33.3] | 0 [0 to 16.7]
  Week 10 | 0 [-16.7 to 33.30] | 0 [0 to 16.7]
  Week 13 | 0 [0 to 16.7] | 0 [-16.7 to 0]
  Week 16 | -16.7 [-33.3 to 0] | 0 [0 to 33.3]
  Week 19 | 0 [0 to 0] | 0 [0 to 0]
  Week 22 | 0 [0 to 0] | 0 [0 to 0]
  Week 25 | 33.3 [33.3 to 33.3] | 0 [0 to 0]
  Week 28 | 0 [0 to 0] | 0 [0 to 0]
  Week 31 | 0 [0 to 0] | 0 [0 to 0]
  Week 34 | 0 [0 to 0] | 0 [0 to 0]
  30 days post last therapy | 0 [-16.7 to 33.3] | 0 [0 to 16.7]

10. Secondary Outcome: HRQoL Questionnaire - EORTC QLQ-C30 Diarrhea
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Diarrhea Scale is scored between 0 and 100 (lower score is better).
Time Frame: Baseline to 30 days after discontinuation (up to 17.6 months)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 42 | 43
units on a scale
  Week 4 | 0 [0 to 0] | 0 [0 to 0]
  Week 7 | 0 [0 to 33.3] | 0 [0 to 0]
  Week 10 | 0 [0 to 0] | 0 [0 to 0]
  Week 13 | 0 [0 to 33.3] | 0 [-33.3 to 0]
  Week 16 | 0 [0 to 0] | 0 [0 to 33.3]
  Week 19 | 0 [0 to 0] | 0 [-16.7 to 0]
  Week 22 | 0 [0 to 0] | 0 [0 to 0]
  Week 25 | 0 [0 to 0] | 0 [0 to 0]
  Week 28 | 0 [0 to 0] | 0 [0 to 0]
  Week 31 | 0 [0 to 0] | 0 [0 to 0]
  Week 34 | 0 [0 to 0] | 0 [0 to 0]
  30 days post last therapy | 0 [0 to 0] | 0 [0 to 33.3]

11. Secondary Outcome: HRQoL Questionnaire - QLQ-BN20 Headache
Description: Health-related quality of life is measured using an EORTC quality of life questionnaire designed specifically for participants with brain tumors (BN-20). Questionnaires may be completed by the participant or with the assistance of the examiner at baseline prior to initiation of study therapy, and then approximately every 8 weeks while on study treatment (prior to discussing treatment response at each visit, whenever possible).
  All single questions are answered using a categorical scale (e.g., 1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much) and linearly transformed to 0 to 100 scales with 1) higher scores for a functional scale representing higher levels of functioning, 2) higher scores for the global health status/quality of life representing higher levels of global health status/quality of life, 3) and higher scores for a symptom scale representing higher level of symptoms. For Headache lower score is better.
Time Frame: Baseline to 30 days after discontinuation (up to 17.6 months)
Population: QLQ-BN20 scores were evaluated in all randomized patients who filled in at least baseline and one post baseline questionnaire. Scores were summarized by means of descriptive statistics. Median differences between treatment groups in change from baseline to every 4 weeks and the inter-quartile range are reported.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 31 | 33
units on a scale
  Week 4 | 0 [-33.3 to 0] | 0 [-33.3 to 0]
  Week 7 | 0 [-33.3 to 33.3] | 0 [0 to 0]
  Week 10 | -33.3 [-66.7 to 33.3] | 0 [-33.3 to 16.7]
  Week 13 | -16.7 [-33.3 to 16.7] | 0 [0 to 16.7]
  Week 16 | -33.3 [-33.3 to -33.3] | 0 [0 to 0]
  Week 19 | 0 [0 to 50.0] | 0 [0 to 0]
  Week 22 | 0 [0 to 0] | 0 [0 to 0]
  Week 25 | 0 [0 to 0] | 0 [0 to 0]
  Week 28 | 0 [0 to 0] | 0 [0 to 0]
  Week 31 | 0 [0 to 0] | 33.3 [33.3 to 33.3]
  Week 34 | 0 [0 to 0] | 66.7 [66.7 to 66.7]
  30 days post last therapy | 0 [-33.3 to 0] | 0 [0 to 33.3]

12. Secondary Outcome: Number of Participants With Adverse Events
Description: A summary of serious adverse events (SAEs) and all other non-serious adverse events is located in the Reported Adverse Event Module.
Time Frame: every 6 weeks (up to 27.2 months)
Population: Safety population of all participants who received at least one dose of study drug. All serious adverse events are reported. Other adverse events are reported with a threshold that they occurred in greater than 5% of patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 54 | 53
Participants
  Adverse Events | 35 | 33
  Serious Adverse Events | 39 | 42

ADVERSE EVENTS:
Arm/Group | Enzastaurin | Placebo
Serious Adverse Events (participants affected / at risk) | 35/54 | 33/53
Other Adverse Events (participants affected / at risk) | 39/54 | 42/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=54) | Placebo (N=53)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 9 (9)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (7)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=54) | Placebo (N=53)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 19 (19) | 8 (9)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 11 (11) | 6 (7)
Chest pain (General disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 6 (6) | 6 (6)
Oedema peripheral (General disorders) | 8 (9) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Oral candidiasis (Infections and infestations) | 2 (2) | 8 (8)
Urine colour abnormal (Investigations) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 4 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 4 (4)
Chromaturia (Renal and urinary disorders) | 6 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days